CLINICAL TRIAL: NCT02013076
Title: Determinants Of Oral Corticosteroid Responsiveness in Wheezing Asthmatic Youth
Acronym: DOORWAY
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Professor Francine Ducharme, Professor, St. Justine's Hospital
Other Study IDs: CHUSJ
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: Asthma; Children; Cohort study; Corticosteroids
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva for cotinine and for DNA and nasopharyngeal samples for viral analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Oral corticosteroids (OCS): All patients receive:
  1. Prednisone or Prednisolone at 1 mg/kg (in 1 site) or 2 mg/kg (in all other sites) (max. 50 mg); if vomiting prednisone/prednisolone: they receive dexamethasone (0.3 mg/kg, max. 10 mg)
  2. 2 to 3 doses of salbutamol within the first hour of therapy according to severity Those with severe exacerbations receive 3 treatments with salbutamol and ipratropium bromide within the initial hour of therapy.

SUMMARY:
The aim of the prospective cohort study is to: (1) document the magnitude of response to oral corticosteroids administered to children presenting to the emergency department with moderate or severe asthma and (2) quantify clinically available potential determinants of the response to corticosteroids, such as age, gender, triggers of the index exacerbation, environmental tobacco smoke (ETS), gene polymorphisms, and their interactions.

DETAILED DESCRIPTION:
The objective of the large multicentre cohort study is to quantify the response to oral corticosteroids in children aged 1 to 17 years presenting to the ED with a moderate or severe asthma exacerbation.

The main outcome is hospital admission within 72 hours of the oral corticosteroid administration.

Secondary outcomes include the change in Pediatric Respiratory Assessment Measure (PRAM), length of active treatment and other markers of response to therapy in the ED as well as markers of recovery over the next 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject will be eligible if he/she:

  1. is aged 1 to 17 years,
  2. has not received any oral, IM or IV corticosteroid within the last 5 days?
  3. Presents to the hospital emergency department with an acute episode of cough, wheezing and/or dyspnea?
  4. Has asthma as defined as one or more of the following 6 criteria:

     (i) prior diagnosis of asthma made by a physician; OR (ii) prior documented episode of acute cough, wheezing and/or dyspnea with significant response to inhaled β2-agonists or to oral corticosteroids; OR (iii) in a child aged <2 years, 3 or more episodes of cough, wheezing and/or dyspnea, including the index visit; OR (iv) previous lung function tests showing significant reversibility post-bronchodilation (≥12% FEV1 or ≥25% Rrs at 4 to 8 Hz); OR (v) a positive provocation test (PC20 ≤8 mg/mL or Provocation Dose (to increase Rrs by 50% or more (PD50) ≤8 mg/mL), OR (vi) the current episode diagnosed or suspected of asthma by the emergency physician?
  5. have moderate or severe airway obstruction, defined as a Paediatric Respiratory Asthma Measure (PRAM) score >3 at baseline,

Exclusion Criteria:

* Patient will be excluded if :

  1. he/she has another chronic respiratory condition (such as bronchopulmonary dysplasia or cystic fibrosis);
  2. there is a reasonable suspicion of bronchiolitis or foreign body aspiration;
  3. he/she has a prior history of hypersensitivity to salbutamol, ipratropium bromide or oral prednisone/prednisolone;
  4. he/she has a relative or absolute contraindication to receiving oral corticosteroids such as recent exposure to varicella or live vaccine in past 14 days,
  5. there is confirmed or suspected pregnancy.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 to 17 years with moderate to severe asthma with Pediatric Respiratory Assessment Measure (PRAM) ≥4.
Sampling Method: Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Hospital admission | 72 hours after oral corticosteroids administration
  Hospital admission or Length of active treatment for 8 or more hours after the oral corticosteroid administration or ED return visit associated with hospital admission within 72 hours after the oral corticosteroid administration or ED return visit associated within 72 hours with length of active treatment for 8 or more hours after the oral corticosteroid administration

SECONDARY OUTCOMES:
Length of active treatment in hospital | 8 hours after oral corticosteroid administration
Meeting the severity criteria for admission | Within 4 hours of oral corticosteroid administration
  Proportion of children with a PRAM score ≥4 within 4 hours of oral corticosteroid administration
PRAM profile in the ED | Within 4 hours of oral corticosteroid administration
  Area under the curve of the PRAM measured hourly for the time of oral corticosteroid (OCS) until 4 hours after OCS
Time to meeting discharge criteria | Within 8 hours of oral corticosteroid administration
  Time until PRAM score ≤ 3
Change in respiratory resistance | Within 4 hours of oral corticosteroid administration
  Change in respiratory resistance between baseline and disposition will be documented on the MasterScreen Impulse Oscillometry (Cardinal Health Canada, Montreal, Canada) using previously described standardized techniques in cooperative children aged ≥3 years. (measured in a subset of individuals)
Unscheduled visits for asthma | Within 7 days of the index ED exacerbation
  unscheduled visits for asthma as reported by parents and confirmed by medical charts.
Symptom score | Within 7 days of the index ED exacerbation
  Area under the curve of symptoms measured daily on the validated Asthma flare-up diary for children
Duration of asthma symptoms | Within 7 days of the index ED exacerbation
  Duration of symptoms measured daily on the validated Asthma flare-up diary for children
Cumulative reliever use | Within 7 days of the index ED exacerbation
  Cumulative number of puffs of reliever medication as recorded daily on the Asthma flare-up diary for children
Duration of use of rescue ß2-agonists | Within 7 days of the index ED exacerbation
  Duration of use of rescue ß2-agonists as recorded on the Asthma flare-up diary for children

OTHER OUTCOMES:
Adverse events | Within 7 days of the index ED exacerbation
  Number of children with vomiting, serious Infection, psychosis, and mood disturbances
Serious Adverse Health Events | Within 7 days of the index ED exacerbation
  Number of children with adverse events requiring hospitalization, prolonged hospitalization, life threatening, other medically important events or associated with significant disability or incapacity

CONTACTS AND LOCATIONS:
Overall Officials: Francine M Ducharme, MD., M.Sc., Principal Investigator — CHU Sainte Justine, University of Montreal
Locations (5):
- Canada (5):
  - Children's Hospital of London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital (MCH), Montreal, Quebec
  - CHU Sainte-Justine (CHUSJ), Montreal, Quebec
  - Centre Hospitaliser de l'Université Laval, Québec, Quebec

REFERENCES:
- [Derived] Tse SM, Krajinovic M, Chauhan BF, Zemek R, Gravel J, Chalut D, Poonai N, Quach C, Laberge S, Ducharme FM; DOORWAY research group of the Pediatric Emergency Research in Canada (PERC) network. Genetic determinants of acute asthma therapy response in children with moderate-to-severe asthma exacerbations. Pediatr Pulmonol. 2019 Apr;54(4):378-385. doi: 10.1002/ppul.24247. Epub 2019 Jan 15. PMID 30644648
- [Derived] Merckx J, Ducharme FM, Martineau C, Zemek R, Gravel J, Chalut D, Poonai N, Quach C; Pediatric Emergency Research Canada (PERC) DOORWAY team. Respiratory Viruses and Treatment Failure in Children With Asthma Exacerbation. Pediatrics. 2018 Jul;142(1):e20174105. doi: 10.1542/peds.2017-4105. Epub 2018 Jun 4. PMID 29866794
- [Derived] Ducharme FM, Zemek R, Chauhan BF, Gravel J, Chalut D, Poonai N, Guertin MC, Quach C, Blondeau L, Laberge S; DOORWAY research group of the Pediatric Emergency Research in Canada (PERC) network. Factors associated with failure of emergency department management in children with acute moderate or severe asthma: a prospective, multicentre, cohort study. Lancet Respir Med. 2016 Dec;4(12):990-998. doi: 10.1016/S2213-2600(16)30160-6. Epub 2016 Jul 20. PMID 27451347
- [Derived] Ducharme FM, Zemek R, Gravel J, Chalut D, Poonai N, Laberge S, Quach C, Krajinovic M, Guimont C, Lemiere C, Guertin MC. Determinants Of Oral corticosteroid Responsiveness in Wheezing Asthmatic Youth (DOORWAY): protocol for a prospective multicentre cohort study of children with acute moderate-to-severe asthma exacerbations. BMJ Open. 2014 Apr 7;4(4):e004699. doi: 10.1136/bmjopen-2013-004699. PMID 24710133